CLINICAL TRIAL: NCT04378413
Title: The Effect of Aquatic and Land Exercises on Pain, Health Related Quality of Life, Kinesiophobia and Disability in Chronic Low Back Pain
Brief Title: Aquatic and Land Exercises in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ayça Aytar TIĞLI, PhD,PT,Assoc.Prof, Baskent University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 62310886-600
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Chronic Low-back Pain
Keywords: Aquatic Exercises; Chronic Low Back Pain,; Land Exercises; Pain,; Functional status
MeSH Terms: conditions — Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Aquatic Exercises on Pain, quality of life (Experimental): Water-based exercise program was conducted in the second group of 15 patients in an indoor swimming pool. Temperature of mineral water was 36 °C. The program included warming up by walking forwards, sideways and backwards through the water in the pool; active range of motion of the joints of the lower extremities; stretching lower extremities; strengthening exercises for hips, knees, arms, elbows and wrists; and cooling down (slow walking, squatting and standing).
  Interventions: Other: exercise
- The Effect of Land Exercises on Pain, Quality of life (Experimental): Land-based exercise program included abdominal and back strengthening exercises.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — exercise for low back pain

SUMMARY:
Aquatic and Land Exercises on Chronic Low Back Pain

DETAILED DESCRIPTION:
The Effect of Aquatic and Land Exercises on Pain, Health Related Quality of Life, Kinesiophobia and Disability in Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

* patients had to be diagnosed with clinical examination and radiological findings of low back pain from at least 6 months.

Exclusion Criteria:

* acute pain

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
pain in low back pain after aqua and land exercises | 4 week
  It is asked to mark pain on a 10 cm scale.Pain was assessed at rest and at movement by using a 10-cm-long visual (0 cm means no pain while 10 cm means worst pain
quality of life after aqua and land exercises | 4 week
  Quality of life was assessed by Short-Form 36 Health Survey (SF-36) High scores indicate good quality of life and low scores represent poor quality of life.

SECONDARY OUTCOMES:
disability in low back paitients after aqua and land exercise | 4 week
  .For disability assessment, the Modified Oswestry Disability İndex was used . According to the sum of scale; 0-4 points were considered as no disability, 5-14 points were mild, 15-24 points were moderate, 25-34 points were serious, and 35-50 points were fully functional inadequacy.
kinesiophobia in low back paitients after aqua and land exercise | 4 week
  The assessment of kinesiophobia was made with the Tampa Scale The fact that the individual got a high score from the questionnaire shows that she has more fear of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayça Aytar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No